CLINICAL TRIAL: NCT00987103
Title: Pharmacokinetic Study to Rectal and Sublingual Administration of Tacrolimus in Future Kidney Transplant Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: A. van de Plas / Hospital Pharmacist, Maastricht University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-2-016
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Organ Transplantation
Keywords: renal transplantation; tacrolimus; pharmacokinetics; rectal; sublingual; rectal administration; sublingual administration
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sublingual - Rectal - Oral (Experimental): Administration order of rank: Sublingual - Rectal - Oral
  Interventions: Drug: Tacrolimus
- Sublingual - Oral - Rectal (Experimental): Administration order of rank: Sublingual - Oral - Rectal
  Interventions: Drug: Tacrolimus
- Oral - Sublingual - Rectal (Experimental): Administration order of rank: Oral - Sublingual - Rectal
  Interventions: Drug: Tacrolimus
- Oral - Rectal - Sublingual (Experimental): Administration order of rank: Oral - Rectal - Sublingual
  Interventions: Drug: Tacrolimus
- Rectal - Sublingual - Oral (Experimental): Administration order of rank: Rectal - Sublingual - Oral
  Interventions: Drug: Tacrolimus
- Rectal - Oral - Sublingual (Experimental): Administration order of rank: Rectal - Oral - Sublingual
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Oral: 0,1 mg/kg Rectal: 15 mg Sublingual: 0,04 mg/kg
  Other Names: Prograft

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of rectal and sublingual administration of tacrolimus and to compare with pharmacokinetics after oral administration of tacrolimus in renal transplant patients before transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will have a kidney transplant patient and will be treated with tacrolimus. As well as hemodialysis patients as well as peritoneal dialysis patients are included.
* Age: 18 - 65 years
* Patient's informed consent

Exclusion Criteria:

* Patients that use drugs that interact with tacrolimus
* Patients that participate in other studies
* Patients that are treated with tacrolimus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Area under the curve, bioavailability, time of maximal concentration, elimination constant | t = 0, ½, 1, 2, 4, 8, 12, 24, 36 and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Johannes van Hooff, Professor, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Hospital, Maastricht, Netherlands